CLINICAL TRIAL: NCT05954949
Title: Detection of Ileoanal Pouch/ Reservoir Adenomas by Routine Chromoendoscopy With Indigocarmine
Brief Title: Detection of Ileoanal Pouch/Reservoir Adenomas
Acronym: DARIAC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jean Christophe Saurin (Other)
Responsible Party: Sponsor-Investigator, Jean Christophe Saurin, Principal Investigator, Medical Doctor, Hôpital Edouard Herriot
Organization: Hôpital Edouard Herriot (Other)
Other Study IDs: SFED 160
Record Dates: First submitted 2023-07-11; First posted 2023-07-20 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Adenomatous Polyps
Keywords: familial adenomatous polyposis; Ileoanal pouch/reservoir; adenomas; chromoendoscopy; indigocarmine; colectomy
MeSH Terms: conditions — Adenomatous Polyps; Adenomatous Polyposis Coli; Adenoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ileoanal pouch adenomas detection assessment: Every patient who needs follow up lower digestive examination for familial adenomatous polyposis after colectomy can join this study with ileal pouch adenomas detection by experienced endoscopist.
  Interventions: Procedure: Adenomas detection rate with the different observation methods

INTERVENTIONS:
Procedure: Adenomas detection rate with the different observation methods — Films performed in white light high definition, NBI and indigo-carmine dye, will be compared blindly to detecte number of adenomas with the different observation methods

SUMMARY:
The detection of adenomas is the basis for the follow-up of patients with familial adenomatous polyposis, after colectomy, with a remnant rectum or an ileal pouch. The optimal method for the adenomas detection is not defined yet. Despite the proven effectiveness of indigo-carmine in different indications dye chromoendoscopy is not used in a consensual way at the international level. The situation of the ileal pouch is specific as adenomas have a usually flat shape and are much more difficult to identify than in the situation of a remnant rectum, even in the situation of > 5 mm adenomas that should be resected.

Our hypothesis is that indigo-carmine can improve adenomas detection, including > 5 mm adenomas, in patients with a an ileal pouch after colectomy improving the effectiveness of surveillance programs and potentially reducing the risk of cancer in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with familial adenomatous polyposis
* Ileo-anal anastomosis with pouch reservoir
* Quality of the final preparation = 3 (excellent) on the studied area
* Films made under optimal conditions for the 3 staining methods

Exclusion Criteria:

* Patient with no familial adenomatous polyposis
* Patient without Ileo-anal anastomosis reservoir
* Insufficient quality of the final preparation <3
* Absence of films made under optimal conditions for the 3 staining methods

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with familial adenomatous polyposis after colectomy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-11 (Estimated)

PRIMARY OUTCOMES:
Average number of ileal pouch/reservoir adenomas | 6 months after colonoscopy
  Average number of ileal pouch/reservoir adenomas detected according to the endoscopic mode (staining or not, virtual or not) based on a paired review of the films with final consensus in case of discordance